CLINICAL TRIAL: NCT04849286
Title: A Phase 1, Open-label, Randomised, Single-centre, Single Oral Dose Study to Determine the Concentration of HTL0016878 in Cerebrospinal Fluid and Plasma in Healthy Male Subjects Following Dosing With HTL0016878 Oral Solution
Brief Title: Measurement of HTL0016878 in Cerebrospinal Fluid
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nxera Pharma UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HTL0016878-103; 2018-002784-26 (EudraCT Number)
Record Dates: First submitted 2021-04-15; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Healthy Subjects
Keywords: Cerebrospinal Fluid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (Experimental): 10 mg dose, CSF sample 2 hours post-dose
  Interventions: Drug: HTL0016878
- Group 2 (Experimental): 10 mg dose, CSF sample 6 hours post-dose
  Interventions: Drug: HTL0016878
- Group 3 (Experimental): 20 mg dose, CSF sample 2 hours post-dose
  Interventions: Drug: HTL0016878
- Group 4 (Experimental): 20 mg dose, CSF sample 6 hours post-dose
  Interventions: Drug: HTL0016878

INTERVENTIONS:
Drug: HTL0016878 — Oral solution

SUMMARY:
A Phase 1, open-label, randomised, single oral dose study to determine the concentration of HTL0016878 in CSF and plasma in healthy male subjects following dosing with HTL0016878 10 mg or 20 mg oral solution

DETAILED DESCRIPTION:
Up to 24 healthy subjects will be enrolled into 4 groups, with 6 subjects per group. Each subject will be randomised to receive a single oral dose of 10 mg or 20 mg HTL0016878 solution and will have a single CSF sample taken via lumbar puncture at either 2 or 6 hours post-dose. Pharmacokinetic blood sampling and safety measures will continue until 24 hours post-dose.

ELIGIBILITY:
Inclusion Criteria:

Subject has a body mass index (BMI) of 18 to 32 kg/m2, inclusive. Healthy as determined by a responsible physician, based on medical evaluation including medical history, physical examination, concomitant medication, vital signs, 12-lead ECG, C-SSRS responses, and clinical laboratory evaluations.

Willingness to comply with requirements or the trial, including contraception requirements.

Able to give fully informed consent.

Exclusion Criteria:

Positive tests for hepatitis B & C, HIV. Clinically relevant history of abnormal physical or mental health. Clinically relevant abnormal laboratory results (including hepatic and renal panels, complete blood count, chemistry or coagulation panel and urinalysis), 12-lead ECG and vital signs, or physical findings.

History of severe adverse reactions or allergies, or history of an anaphylactic reaction to prescription or non-prescription medication or food.

Drug or alcohol abuse. Smoking. Use of medication that inhibits CYP2D6. Participation in other clinical trials of unlicensed medicines in the previous 3 months. Loss of more than 400 mL blood in the previous 3 months. Vital signs, QTcF interval or laboratory values outside the acceptable range. Predicted poor and intermediate CYP2D6 metabolisers. Clinically relevant abnormal findings at the screening assessment. History of epilepsy or seizures. Clinically relevant abnormal medical history or concurrent medical condition disease associated with cognitive impairment and/or psychosis. History of suicidal thoughts or ideation, or any history of insomnia. Use of tobacco and/or nicotine containing products within 90 days of dosing. Habitual and heavy consumption of caffeinated beverages. Consumption of cranberry, pomegranate, star fruit, grapefruit, pomelos, exotic citrus fruits or Seville oranges (including marmalade and juices made from these fruits) within 3 days before admission. Objection by General Practitioner

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2018-12-07 (Actual); Study Completion 2018-12-07 (Actual)

PRIMARY OUTCOMES:
Concentration of HTL0016878 in CSF | 2 hours
  Pharmacokinetics
Concentration of HTL0016878 in CSF | 6 hours
  Pharmacokinetics
Concentration of HTL0016878 in plasma Cmax | 0-24 hours
  Pharmacokinetics
Concentration of HTL0016878 in plasma AUC | 0-24 hours
  Pharmacokinetics

SECONDARY OUTCOMES:
Treatment Emergent Adverse events | Baseline up to 10 days post-dose
  Safety and Tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- MAC Clinical Research, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No